CLINICAL TRIAL: NCT04630535
Title: Obstructive Sleep Apnea as a Remote Ischemic Preconditioning in Patients Scheduled for Aorto-bifemoral Bypass Surgery
Brief Title: OSA as a Remote Ischemic Preconditioning in Vascular Surgery
Status: Recruiting | Type: Observational
Sponsor: St. Anne's University Hospital Brno, Czech Republic (Other)
Collaborators: Masaryk University (Other)
Responsible Party: Principal Investigator, Ivan Cundrle, Principal Investigator, St. Anne's University Hospital Brno, Czech Republic
Other Study IDs: IIT/2019/25
Record Dates: First submitted 2020-11-04; First posted 2020-11-16 (Actual); Last update posted 2025-05-15 (Actual); Status verified 2025-05

CONDITIONS: Obstructive Sleep Apnea; Vascular Aneurysm; Ischemia Reperfusion Injury
Keywords: remote preconditioning
MeSH Terms: conditions — Sleep Apnea, Obstructive; Reperfusion Injury

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — frozen blood plasma
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Obstructive Sleep Apnea: Pacient with OSA (AHI≥5) undergoing aorto-bifemoral bypass
  Interventions: Procedure: aorto-bifemoral bypass surgery
- Without Obstructive Sleep Apnea: Patinets without OSA undergoing aorto-bifemoral bypass
  Interventions: Procedure: aorto-bifemoral bypass surgery

INTERVENTIONS:
Procedure: aorto-bifemoral bypass surgery — aorto-bifemoral bypass surgery (Leriche syndrom, elective AAA repair)

SUMMARY:
Ischemia and reperfusion (I/R) injury during abdominal aortic aneurysm (AAA) repair is inevitable and may lead to postoperative multi-organ failure. Remote ischemic preconditioning (short periods of ischemia in anticipation of longer period of ischemia) may act protectively against ischemia.

Studies of ischemic preconditioning in patients with AAA are conflicting. Obstructive sleep apnea (OSA) is a sleep disordered breathing syndrome which may have a protective effect against ischemia.

The investigators hypothesize that I/R injury will be less pronounced in patients who have OSA and that the extent of I/R injury will inversely correlate with OSA severity. Accordingly, the aim of this study is to compare postoperative complications and markers of I/R in patients undergoing elective AAA repair who do and do not have OSA.

DETAILED DESCRIPTION:
Patients. Consecutive patients scheduled for elective aortobifemoral bypass (AAA and Leriche syndrome patients) will be recruited for this prospective, observational study.

Polygraphy (PG). PG measurements will be done two nights before surgery using the Embletta system (Embla - Embletta MPR PG Sleep Data Recording System).

STOP-BANG, Epworth questionnaire. Both questionnaires will be done the same day as polygraphy

Cardiovascular complications will be assessed from the first 30 post-operative days Pulmonary complications will be assessed from the first 30 post-operative days

Specific markers of I/R. T0 - before anesthesia induction T1 - 3 hrs after aorta de-clamping T2 - 12 hrs after aorta de-clamping T3 - 24 hrs after aorta de-clamping T4 - on the fifth post-operative day

ELIGIBILITY:
Inclusion Criteria:

* patients scheduled for elective aorto-bifemoral bypass (AAA and Leriche syndrome patients)

Exclusion Criteria:

* emergent surgery
* aorto-bifemoral bypass using deep vein graft
* re-operations
* known OSA with CPAP treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: consecutive patients scheduled for elective aorto-bifemoral bypass (AAA and Leriche syndrome patients)
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2020-11-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Change of I/R injury markers | T0 - before anesthesia induction; T1 - 3 hrs after aorta de-clamping; T2 - 12 hrs after aorta de-clamping; T3 - 24 hrs after aorta de-clamping; T4 - on the fifth post-operative day
  Plasma Total Antioxidant Capacity and Reactive Oxygen Species Concentration

SECONDARY OUTCOMES:
post-operative complications | up to 30 post-operative days
  cardiovascular and pulmonary post-operative complications

CONTACTS AND LOCATIONS:
Overall Officials: Ivan Cundrle, M.D., Ph.D., Principal Investigator — St. Anne's University Hospital in Brno
Locations (1):
- St. Anne's University Hospital Brno, Brno, Czech Republic, Czechia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Katseni K, Chalkias A, Kotsis T, Dafnios N, Arapoglou V, Kaparos G, Logothetis E, Iacovidou N, Karvouni E, Katsenis K. The Effect of Perioperative Ischemia and Reperfusion on Multiorgan Dysfunction following Abdominal Aortic Aneurysm Repair. Biomed Res Int. 2015;2015:598980. doi: 10.1155/2015/598980. Epub 2015 Dec 21. PMID 26798637
- [Background] Murry CE, Jennings RB, Reimer KA. Preconditioning with ischemia: a delay of lethal cell injury in ischemic myocardium. Circulation. 1986 Nov;74(5):1124-36. doi: 10.1161/01.cir.74.5.1124. PMID 3769170
- [Background] Walsh SR, Boyle JR, Tang TY, Sadat U, Cooper DG, Lapsley M, Norden AG, Varty K, Hayes PD, Gaunt ME. Remote ischemic preconditioning for renal and cardiac protection during endovascular aneurysm repair: a randomized controlled trial. J Endovasc Ther. 2009 Dec;16(6):680-9. doi: 10.1583/09-2817.1. PMID 19995115
- [Background] Walsh SR, Sadat U, Boyle JR, Tang TY, Lapsley M, Norden AG, Gaunt ME. Remote ischemic preconditioning for renal protection during elective open infrarenal abdominal aortic aneurysm repair: randomized controlled trial. Vasc Endovascular Surg. 2010 Jul;44(5):334-40. doi: 10.1177/1538574410370788. Epub 2010 May 18. PMID 20484066
- [Background] Li C, Li YS, Xu M, Wen SH, Yao X, Wu Y, Huang CY, Huang WQ, Liu KX. Limb remote ischemic preconditioning for intestinal and pulmonary protection during elective open infrarenal abdominal aortic aneurysm repair: a randomized controlled trial. Anesthesiology. 2013 Apr;118(4):842-52. doi: 10.1097/ALN.0b013e3182850da5. PMID 23353795
- [Background] Murphy N, Vijayan A, Frohlich S, O'Farrell F, Barry M, Sheehan S, Boylan J, Conlon N. Remote ischemic preconditioning does not affect the incidence of acute kidney injury after elective abdominal aortic aneurysm repair. J Cardiothorac Vasc Anesth. 2014 Oct;28(5):1285-92. doi: 10.1053/j.jvca.2014.04.018. PMID 25281045
- [Background] Healy DA, Boyle E, McCartan D, Bourke M, Medani M, Ferguson J, Yagoub H, Bashar K, O'Donnell M, Newell J, Canning C, McMonagle M, Dowdall J, Cross S, O'Daly S, Manning B, Fulton G, Kavanagh EG, Burke P, Grace PA, Moloney MC, Walsh SR; Preconditioning Shields Against Vascular Events in Surgery (Preconditioning SAVES) Trial Group. A MultiCenter Pilot Randomized Controlled Trial of Remote Ischemic Preconditioning in Major Vascular Surgery. Vasc Endovascular Surg. 2015 Nov;49(8):220-7. doi: 10.1177/1538574415614404. Epub 2015 Nov 16. PMID 26574485
- [Background] Garcia S, Rector TS, Zakharova M, Herrmann RR, Adabag S, Bertog S, Sandoval Y, Santilli S, Brilakis ES, McFalls EO. Cardiac Remote Ischemic Preconditioning Prior to Elective Vascular Surgery (CRIPES): A Prospective, Randomized, Sham-Controlled Phase II Clinical Trial. J Am Heart Assoc. 2016 Sep 29;5(10):e003916. doi: 10.1161/JAHA.116.003916. PMID 27688236
- [Background] Thomas KN, Cotter JD, Williams MJ, van Rij AM. Repeated Episodes of Remote Ischemic Preconditioning for the Prevention of Myocardial Injury in Vascular Surgery. Vasc Endovascular Surg. 2016 Apr;50(3):140-6. doi: 10.1177/1538574416639150. Epub 2016 Apr 12. PMID 27075990
- [Background] Mouton R, Pollock J, Soar J, Mitchell DC, Rogers CA. Remote ischaemic preconditioning versus sham procedure for abdominal aortic aneurysm repair: an external feasibility randomized controlled trial. Trials. 2015 Aug 25;16:377. doi: 10.1186/s13063-015-0899-3. PMID 26303818
- [Background] De Freitas S, Hicks CW, Mouton R, Garcia S, Healy D, Connolly C, Thomas KN, Walsh SR. Effects of Ischemic Preconditioning on Abdominal Aortic Aneurysm Repair: A Systematic Review and Meta-analysis. J Surg Res. 2019 Mar;235:340-349. doi: 10.1016/j.jss.2018.09.049. Epub 2018 Nov 13. PMID 30691816
- [Background] Sanchez-de-la-Torre A, Soler X, Barbe F, Flores M, Maisel A, Malhotra A, Rue M, Bertran S, Aldoma A, Worner F, Valls J, Lee CH, Turino C, Galera E, de Batlle J, Sanchez-de-la-Torre M; Spanish Sleep Network( *). Cardiac Troponin Values in Patients With Acute Coronary Syndrome and Sleep Apnea: A Pilot Study. Chest. 2018 Feb;153(2):329-338. doi: 10.1016/j.chest.2017.06.046. Epub 2017 Jul 20. PMID 28736306
- [Background] Shah N, Redline S, Yaggi HK, Wu R, Zhao CG, Ostfeld R, Menegus M, Tracy D, Brush E, Appel WD, Kaplan RC. Obstructive sleep apnea and acute myocardial infarction severity: ischemic preconditioning? Sleep Breath. 2013 May;17(2):819-26. doi: 10.1007/s11325-012-0770-7. Epub 2012 Oct 23. PMID 23090861